CLINICAL TRIAL: NCT03707600
Title: State and Trait Mediated Response to TMS in Substance Use Disorder
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI closing his lab
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 999918148; 18-DA-N148
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2019-10

CONDITIONS: Nicotine Dependence
Keywords: Nicotine Abstinence; Metaplasticity; Nicotine; Functional Magnetic Resonance Imaging (fMRI); Transcranial Magnetic Stimulation (TMS)
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham (Sham Comparator): The sham coil setting is designed to mimic the auditory artifact and scalp sensations evoked by the real coil without stimulating the brain.
  Interventions: Device: TMS
- TMS (Active Comparator): Active TMS
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — MagVenture MagPro 100 with MagOption (MagVenture Inc, Alpharetta, GA) machine equipped with a figure-8 coil.

SUMMARY:
OBJECTIVES: The current protocol seeks to develop brain-based intermediate phenotypes of response to transcranial magnetic stimulation (TMS) in chronic substance use disorder (SUD). To date the field has relied on subjective reports, behavioral performance, and long-term clinical outcomes as primary measures of TMS efficacy. While certainly ecologically valid, these observable behaviors lack the sensitivity necessary to fully quantify the effects (or lack thereof) across both individual participants and TMS intervention protocols.

This proposed within-subjects design seeks to leverage differences in metaplasticity that is, the context in which stimulation occurs-by studying the response to stimulation in both sated and abstinent states. It is predicted these state manipulations will potentiate response to TMS. When a disruptive allostatic load like chronic nicotine exposure or acute abstinence is placed on the brain, the underlying network becomes less stable and thus more susceptible to TMS intervention. For SUD in general and tobacco use disorder (TUD) in particular, this state dependence of TMS response is a potentially valuable tool to improve a given intervention s clinical efficacy.

STUDY POPULATION: Physically and psychiatrically healthy smokers will be recruited. A comparison group of non-smokers will be concurrently enrolled. We estimate we will require n=51/group of completers to have sufficient power to develop the intermediate phenotypes of TMS.

DESIGN: The protocol is a two group, between/within subject, fully counterbalanced design. The between-subjects factor is GROUP (smoker/non-smoker) and the within-subjects factor for each GROUP is TMS CONDITION (active/sham). Additionally, and for the smoker group, nicotine STATE (sated/abstinent) is a nested within-subjects factor. Each group will receive single sessions of active and sham intermittent theta burst stimulation to left dorsal lateral prefrontal cortex, followed immediately by an MRI scan to characterize the acute neurobiological response to stimulation. Smokers will repeat these procedures both during smoking satiety and following an ~48-hour period nicotine abstinence.

OUTCOMES PARAMETERS: In addition to subjective and behavioral task performance changes associated with TMS intervention, changes in MRI BOLD signal will be used to characterize the neurobiological response to TMS intervention across groups and states. Taken together, the development of brain-based markers of TMS response may thus improve both our mechanistic understanding of the causal dysfunctions of TUD as well as the potential efficacy of these interventions longer term to address the relevant clinical characteristics of the disease and ultimately improve treatment outcomes.

DETAILED DESCRIPTION:
OBJECTIVES: The current protocol seeks to develop brain-based intermediate phenotypes of response to transcranial magnetic stimulation (TMS) in chronic substance use disorder (SUD). To date the field has relied on subjective reports, behavioral performance, and long-term clinical outcomes as primary measures of TMS efficacy. While certainly ecologically valid, these observable behaviors lack the sensitivity necessary to fully quantify the effects (or lack thereof) across both individual participants and TMS intervention protocols.

This proposed within-subjects design seeks to leverage differences in metaplasticity that is, the context in which stimulation occurs-by studying the response to stimulation in both sated and abstinent states. It is predicted these state manipulations will potentiate response to TMS. When a disruptive allostatic load like chronic nicotine exposure or acute abstinence is placed on the brain, the underlying network becomes less stable and thus more susceptible to TMS intervention. For SUD in general and tobacco use disorder (TUD) in particular, this state dependence of TMS response is a potentially valuable tool to improve a given intervention s clinical efficacy.

STUDY POPULATION: Physically and psychiatrically healthy smokers will be recruited. A comparison group of non-smokers will be concurrently enrolled. We estimate we will require n=51/group of completers to have sufficient power to develop the intermediate phenotypes of TMS.

DESIGN: The protocol is a two group, between/within subject, fully counterbalanced design. The between-subjects factor is GROUP (smoker/non-smoker) and the within-subjects factor for each GROUP is TMS CONDITION (active/sham). Additionally, and for the smoker group, nicotine STATE (sated/abstinent) is a nested within-subjects factor. Each group will receive single sessions of active and sham intermittent theta burst stimulation to left dorsal lateral prefrontal cortex, followed immediately by an MRI scan to characterize the acute neurobiological response to stimulation. Smokers will repeat these procedures both during smoking satiety and following an ~48-hour period nicotine abstinence.

OUTCOMES PARAMETERS: In addition to subjective and behavioral task performance changes associated with TMS intervention, changes in MRI BOLD signal will be used to characterize the neurobiological response to TMS intervention across groups and states. Taken together, the development of brain-based markers of TMS response may thus improve both our mechanistic understanding of the causal dysfunctions of TUD as well as the potential efficacy of these interventions longer term to address the relevant clinical characteristics of the disease and ultimately improve treatment outcomes.

ELIGIBILITY:
* INCLUSION CRITERIA (MAIN STUDY):

All participants must:

* Be between the ages of 18-60. Justification: Many neural processes change with age, and these changes could introduce unwanted variability in both behavioral and MRI signals. In addition, the risk of difficult-to-detect medical abnormalities such as silent cerebral infarcts increase with age. Assessment tools: History. Government- issued forms of identification (e.g. driver s license, birth certificate) will be required when participant appears to be out of age range.
* Be in good health. Justification: Many illnesses may alter fMRI signals as well as cognitive processes and neural functioning. Assessment tools: Medical Assessment, Medical History and Physical Examination. Medical assessments include: Vital Signs, EKG, oral HIV test, height/weight measurements, urinalysis and blood sample. Tests on the blood sample include CBC, complete metabolic profile, TSH, ESR, STS and HIV (if needed to confirm a positive salivary test for HIV). The following individual laboratory results will independently disqualify individuals: Cholesterol greater than 250 mg/dl, Hemoglobin less than 10.5 g/dl, WBC less than 2400/ (Micro)l, LFTs less than 3 times upper normal, HCG positive, Casual serum glucose less than 200 mg/dl, Urine protein less than 1+. The MAI will retain discretion to exclude at less extreme values, depending on the clinical presentation. (Serum glucose over 140 mg/dl will be followed up with a fasting serum glucose assessment. Those with fasting glucose below 100 mg/dl may be considered for the protocol. Others will be rejected and referred for work-up.) Liver function will be evaluated with aspartate aminotransferase (AST) and alanine transaminase (ALT). A greater than 3 times upper normal limit for AST or ALT will disqualify individuals. MAI will make the final judgment on any questionable lab results.
* Be right-handed. Justification: Using right-handed individuals will reduce variability in BOLD MRI data. Assessment tool: Edinburgh Handedness Inventory.
* Be able to abstain from alcohol and other substances 24hrs and caffeine for 12 hours before each of the imaging sessions. Justification: Alcohol and caffeine (among other substances) modulate neural functioning in a way that would complicate data interpretation. Assessment tools: Self-report, urine drug screen and breathalyzer.
* For smoker group, must have a urine cotinine level of greater than 4 as measured by a semi-quantitative in vitro diagnostic (e.g., NicAlert) and have been smoking a regular combustible tobacco product consistently for at least one year. Based on the correlation between self-reported cpd/FTND and urine cotinine levels, a single inclusion criterion will be easier to manage and provide adequate characterization of dependent smokers. Urine cotinine level provides a biomarker that does not rely on self-report/memory. Quit attempts will be assessed via clinical interview and judgment. Justification: The present protocol is interested in neurobiological mechanisms that underlie nicotine dependence-induced plasticity, and is thus contingent on the presence of nicotine dependence. Assessment tools: Self-report, NicAlert of 4 or higher (or other nicotine/cotinine lab test equivalent to 200ng/ml cotinine concentration)
* For the smoker group, must be willing to attempt an acute abstinence period lasting approximately 48 hours on 2 separate occasions. Justification: We aim to look at the response to stimulation in both drug sated and abstinent states in smokers. Assessment tool: Self-report.
* For the non-smoking control group, less than 20 cigarettes lifetime, no cigarette or other nicotine product in past year and no history of daily use of any other nicotine products for > 2 weeks. Justification: Minimal cigarette exposure in the control group is required to assess differences between healthy control and the smoker groups. Assessment tools: Self-report, NicAlert of less than or equal 2, CO less than 6 or MAI discretion if there is a reasonable planation for high CO exposure.

EXCLUSION CRITERIA (MAIN STUDY):

* Current or personal history of cerebrovascular or neurological illnesses including, but not limited to, seizure disorders, frequent migraines or on prophylaxis, multiple sclerosis, movement disorders, history of significant head trauma, or CNS tumor. Current or personal history of any neurological disorders that would increase seizure risk from iTBS such as stroke, brain lesions, previous neurosurgery, any history of seizure or fainting episode of unknown cause, or head trauma resulting in loss of consciousness, lasting over 30 minutes or with sequela lasting longer than three months, regardless of loss of consciousness. Justification: Cerebrovascular and neurological conditions may alter blood flow, CNS function, the fMRI signal and other autonomic signals. Additionally, neurological disorders such as stroke, vascular lesions or head trauma can lower the seizure threshold and are therefore contra-indications for iTBS. Fainting episodes or syncope of unknown cause could indicate an undiagnosed condition associated with seizures. Assessment tools: TMS Safety Screen and Medical History and Physical Exam. The MAI who will also retain discretion to exclude based on a history of neurological illness that may compromise data integrity.
* First-degree family history of any neurological disorder with a potentially hereditary basis, including migraines, epilepsy, or multiple sclerosis. Justification: Neurological disorders can lower the seizure threshold and are therefore contra-indications for iTBS. First -degree family history of certain neurological disorder with a hereditary component increases the risk of the participant having an undiagnosed conditi n that is associated with lowered seizure threshold. Assessment tools: TMS Safety Screen and Medical History.
* Implantable defibrillator, implanted medication pumps, cardiac pacemaker, neurostimulator, some artificial joints, metal pins, surgical clips, intracardiac lines, or acute unstable cardiac disease with intracranial implants (e.g. aneurysm clips, shunts, stimulators, cochlear implants or electrodes) or any other implant or metal object in the body that precludes MRI scanning or iTBS administrations. Justification: certain metal in the body is a contra-indication for MRI scanning and iTBS administration, which involves exposure to a relatively strong static magnetic field that can move magnetic material not securely bound and rapidly alternating magnetic fields that can generate heat and current in metal contained in the body. Assessment tools: TMS Safety Screen, MRI Safety Screen and Medical History.
* Are not suitable to undergo an fMRI experiment due to body morphology or claustrophobia. Justification: MR scanning is one of the primary measurement tools used in the protocol. Assessment tools: MRI Safety Screen, Medical History. Prospective participants will be questioned about symptoms of claustrophobia and may be placed in the mock scanner during screening to assess for possible difficulty tolerating the confinement of the scanner and for ability to fit into the scanner. Noise-induced hearing loss or tinnitus. Justification: individuals with noise-induced hearing problems may be particularly vulnerable to the acoustic noise generated by iTBS equipment and MRI (even with the use of sound attenuation ear plugs). Assessment tools: TMS Safety Screen, MRI Safety Screen, Medical History.
* Current use (any use in the past 4 weeks, daily use for more than a week within the past 6 months) of any substances (excluding alcohol, see criteria 9), investigational drug or of any medications with psychotropic, anti- or pro-convulsive action, or anti coagulants. This will be determined at the discretion of the MAI. Justification: the use of certain medications or drugs can lower seizure threshold during use or withdrawal and is therefore contra-indicated for iTBS. Assessment tools: Medical History, urine toxicology analysis for the presence of a broad range of prescription and non-prescription drugs. Lifetime history of schizophrenia, bipolar disorder, mania, or hypomania. Justification: The population of interest here is a healthy population with no psychiatric disorders other than tobacco use disorders. In participants with bipolar disorder, mania or hypomania, there is a small chance that iTBS can trigger (hypo)manic symptoms. Assessment tools: M.I.N.I. Potential diagnoses will be further evaluated by a counselor.
* Current major psychiatric disorders to include, but not limited to, mood, anxiety, psychotic disorders, or substance-induced psychiatric disorders, or any current suicidal ideations or currently under antidepressant or antipsychotic medication treatment. The MAI will reserve the right to exclude on the basis of psychiatric history not explicitly described in this criterion. Justification: Psychiatric disorders involve the central neural system (CNS) and, therefore, can be expected to alter the fMRI measures being used in this study. Assessment tools: M.I.N.I., Beck Depression Inventory, Beck Anxiety Inventory, Adult ADHD Self-Report Scales and clinical terview confirmation by clinician.
* Meet current DSM-5 criteria for moderate to severe substance use disorder, for alcohol or any drug (except nicotine for the smoker group). Past substance use disorder (SUD) is acceptable based on MAI determination. Those with past SUD of substances other than alcohol or marijuana may not have any current use (past 6 months) of the substance on which they were dependent. Individuals with past SUD of either alcohol or marijuana who report current use of the previously dependent substance may be included provided they do not currently meet withdrawal criteria. Justification: SUD of other substances (drugs or alcohol) may result in unique CNS deficits that could confound results and introduce excessive variance. Assessment tools: The Mini International Neuropsychiatric Interview (M.I.N.I) and clinical SUD assessment, Drug Use Survey, Addiction Severity Index. A positive drug test for marijuana will not be exclusionary as long as participants, based on self- report, have not used in the 24hrs preceding the imaging visits. In the event of a positive drug test for marijuana, self-reports of current marijuana use will be used to differentiate intermittent/infrequent from chronic/frequent users.
* History of myocardial infarction, angina, congestive heart failure, cardiomyopathy, stroke or transient ischemic attack, mitral valve prolapse, or any heart condition currently under medical care. Justification: the risk of iTBS for individuals with a heart condition is unknown, further such conditions may alter blood flow, the fMRI signal and other autonomic signals. These conditions are also likely to add considerable additional variability to the data. Assessment tools: physical assessment, EKG, medical history.
* Women who are pregnant, sexually active and not using an acceptable form of birth control. Justification: study procedures used in the current protocol (MRI, iTBS) may complicate pregnancy. Assessment tools: Urine and/or serum pregnancy tests, and clinical interview. Urine pregnancy tests will also be conducted at the beginning of each imaging visit.
* Participation in any NIBS session (excluding the current protocol) less than two weeks ago. No NIBS exposure for treatment purposes in the last 6 months. Justification: in order to avoid possible carry-over effects from previous exposure to NIBS prior to participation in the proposed intervention, we will not enroll participants who have received any NIBS in the two weeks preceding enrollment or treatment with NIBS modality with the last 6 months preceding enrollment. Assessment tools: TMS safety screen.
* Cognitively impaired or learning disabled. Justification: Cognitive impairment and learning disabilities may be associated with altered brain functioning in regions recruited during laboratory task performance. Cognitive impairment may affect one s ability to give informed consent. Assessment tool: Medical History and Wechsler Abbreviated Scale of Intelligence (WASI). IQ estimate must be 80 or over.
* Have coagulopathies, history of, current superficial, or deep vein thrombosis, musculoskeletal abnormalities restricting an individual s ability to lie flat for extended periods of time. Justification: MR scanning sessions require participants to lie flat on their backs and remain perfectly still for approximately two hours. Therefore, conditions that would make that difficult (e.g. chronic back pain, significant scoliosis) or dangerous (e.g. familial hypercoagulability syndrome, history of thrombosis) will be exclusionary. Assessment tools: History and physical examination by a qualified IRP clinician, supplemented with a trial of lying in the mock scanner to ssess comfort issues.
* Regularly use any prescription (e.g., antidepressants, benzodiazepines, antipsychotics, anticonvulsants, barbiturates), over-the-counter (e.g., cold medicine) or herbal medication (e.g., Kava, Gingko biloba, St. John s wort) that may alter CNS function, cardiovascular function, or neuronal-vascular coupling. Justification: The use of these substances may alter the fMRI signal and/or neural functions of interest in the current study. Assessment tools: History and comprehensive urine drug screening to detect antidepressants, benzodiazepines, antipsychotics, anticonvulsants, and barbiturates.

INCLUSION CRITERIA (PROTOCOL TRIANING):

Participants must:

* Be Right-handed.

  * Justification: Differences in hemispheric dominance could confound iTBS administration and MRI measurements.
  * Screening tool: Self-report.
* Be in good health.

  * Justification: Many illnesses may increase likelihood of TMS ...

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Subjective and behavioral task report and changes in MRI BOLD signal | Each TMS/MRI visit
  changes in MRI BOLD signal

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Stein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States